CLINICAL TRIAL: NCT03048019
Title: Comparison of Pharmacodynamic Effects of Tirofiban vs. Cangrelor in N-STEMI Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Antiplatelet Effects of Tirofiban vs. Cangrelor N-STEMI Patients Undergoing Percutaneous Coronary Intervention
Status: Terminated | Type: Observational
Why Stopped: study terminated per PI
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Other Study IDs: 17-2617
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Non-ST Elevation Myocardial Infarction (NSTEMI)
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Tirofiban; cangrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tirofiban Therapy: patients randomized to tirofiban therapy
  Interventions: Drug: Tirofiban
- Cangrelor Therapy: patients randomized to cangrelor therapy
  Interventions: Drug: Cangrelor

INTERVENTIONS:
Drug: Tirofiban — Patients will receive Tirofiban during the PCI procedure
  Other Names: Aggrastat
  Groups: Tirofiban Therapy
Drug: Cangrelor — Patients will receive Cangrelor during the PCI procedure
  Other Names: Kengreal
  Groups: Cangrelor Therapy

SUMMARY:
Immediate potent inhibition of platelet function is critical for the prevention of periprocedural ischemic event occurrences in high risk N-ST segment elevation myocardial infarction (NSTEMI) in patients undergoing percutaneous coronary intervention (PCI). Currently, dual antiplatelet therapy with aspirin and an oral P2Y12 receptor blocker (with loading doses) is widely used for PCI. However, immediate, potent and reversible inhibition of platelet aggregation is not possible even with the newer oral agents, prasugrel and ticagrelor. Therefore, an intravenously administered GPIIb/IIIa receptor inhibitor (tirofiban) or P2Y12 receptor blocker (cangrelor) with fast onset and offset of actions will provide more desired antiplatelet effects in the setting of PCI. This study will measure and compare the anti-platelet effects of Tirofiban and Cangrelor in patients presenting with N-STEMI and undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

1. NSTEMI meeting the following criteria:

1. Patients 18 years of age or older with one or more of the following symptoms:

   * new ST-segment depression or transient elevation of at least 1 mm
   * elevations in troponin I, troponin T, or creatine kinase MB levels above ULN
2. Eligible for ticagrelor, cangrelor, aspirin, UFH, and GP IIb/IIIa inhibitor treatment.
3. Admitted at cardiac catheterization laboratory hospital or associated facility.
4. Competent mental condition to provide informed consent.

Exclusion Criteria:

1. Unstable angina, STEMI
2. Cardiogenic shock
3. Refractory ventricular arrhythmias
4. New York Heart Association class IV congestive heart failure
5. Cardiac arrest within 1 week of study entry
6. History of hemorrhagic or ischemic stroke, TIA, sub-arachnoid hemorrhage or intracranial neoplasm, arteriovenous malformation, or aneurysm
7. Fibrinolytic therapy within 48 hours of study entry
8. Active pathological bleeding or history of bleeding diathesis
9. Severe hepatic insufficiency
10. Current peptic ulceration
11. Increased bleeding risk, per investigator judgment
12. Known anemia (hematocrit<25%)/thrombocytopenia (platelet count < 100,000mm3)
13. Surgery within 4 weeks before study entry or planned surgery within 2 months after study entry
14. Any P2Y12 receptor inhibitor or GP IIb/IIIa inhibitor within 7 days of study entry
15. Receiving warfarin or other coumadin derivatives or NOACs within the last 10 days with an INR >1.5 secs or planned use during the hospitalization period
16. Contraindication to the use of ticagrelor and/or aspirin
17. Receiving or will receive oral anticoagulation or other oral antiplatelet therapy (except aspirin) that cannot be safely discontinued within the next 3 months
18. Receiving daily NSAIDs or COX2 inhibitors that cannot be discontinued or anticipated to require >2 weeks of daily NSAIDs or COX2 inhibitors during study
19. Investigational drug in last 30 days or presently enrolled in drug/device study
20. Women of childbearing potential (post-menopausal women can be enrolled if at least 1 year of amenorrhea or surgically sterile)
21. Condition associated with poor treatment compliance (e.g., alcoholism, mental illness, or drug dependence)
22. Inability to provide written informed consent and to understand the full meaning of the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will consist of NSTEMI patients undergoing percutaneous coronary intervention (PCI): 30 patients each will be treated with tirofiban or cangrelor (total n=60).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gurbel, MD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Health Care System, Falls Church, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 participants were enrolled. 18 participants were screen failures as they did not require coronary stenting. 10 participants were assigned treatment.
Period: Overall Study
Arm/Group | Tirofiban Therapy | Cangrelor Therapy
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tirofiban Therapy | Cangrelor Therapy | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (12.1) | 57.3 (12.2) | 57.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Thrombin Receptor Activator Peptide (TRAP) Induced Platelet Aggregation (%)
Description: Assessment of platelet aggregation (%) in response to 10uM thrombin receptor activator peptide. Normal reference range is 60-100% aggregation.
Time Frame: 30 minutes post-start of the infusion
Measure: Mean (Standard Deviation); unit: % aggregation
Arm/Group | Tirofiban Therapy | Cangrelor Therapy
Number analyzed (Participants) | 5 | 5
% aggregation | 42.5 (10.2) | 71.2 (6.9)

2. Secondary Outcome: Adenosine Diphosphate (ADP) Induced Platelet Aggregation (%)
Description: Assessment of platelet aggregation (%) in response to 20uM ADP at baseline and serially following tirofiban or cangrelor infusion. Normal reference range is 60-100% aggregation.
Time Frame: 30 minutes post-start of the infusion
Measure: Mean (Standard Deviation); unit: % aggregation
Arm/Group | Tirofiban Therapy | Cangrelor Therapy
Number analyzed (Participants) | 5 | 5
% aggregation | 3.3 (3.1) | 39.4 (13.1)

3. Secondary Outcome: Thrombin Induced Platelet-fibrin Clot Strength (mm)
Description: Assessment of thrombin induced platelet-fibrin clot strength (mm) by thromboelastography (TEG6S). Normal reference range is 55-68 mm
Time Frame: 30 minutes post-start of the infusion
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tirofiban Therapy | Cangrelor Therapy
Number analyzed (Participants) | 5 | 5
mm | 63.9 (2.7) | 62.3 (3.6)

4. Secondary Outcome: Shear-induced Thrombus Formation (AUC)
Description: Real time evaluation of shear-induced thrombus formation using novel RUO T-TAS plus system. AUC is calculated as time to reach 60 kPa
Time Frame: 30 minutes after the end of the infusion.
Measure: Mean (Standard Deviation); unit: kPa*min
Arm/Group | Tirofiban Therapy | Cangrelor Therapy
Number analyzed (Participants) | 5 | 5
kPa*min | 14.1 (13.7) | 1004 (884)

ADVERSE EVENTS:
Time Frame: Up to 48 hours after discharge
Arm/Group | Tirofiban Therapy | Cangrelor Therapy
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tirofiban Therapy (N=5) | Cangrelor Therapy (N=5)
Bleeding (Surgical and medical procedures) | 1 (1) | 0 (0) — Type 2 BARC Bleeding
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tirofiban Therapy (N=5) | Cangrelor Therapy (N=5)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT03048019/Prot_SAP_000.pdf